CLINICAL TRIAL: NCT02848040
Title: The Role of Faecal Bile Acids in the Management of Bile Acid Diarrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016GAS85
Record Dates: First submitted 2016-07-20; First posted 2016-07-28 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Bowel Diseases
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): All patients will receive the same interventions. Single are only
  Interventions: Other: IDK Bile Acids

INTERVENTIONS:
Other: IDK Bile Acids — colourimetric in-vitro laboratory diagnostic test

SUMMARY:
Bile acid malabsorption (BAM), a common cause of diarrhoea, affects 1 million people in the UK, but is often misdiagnosed as irritable bowel syndrome or goes unrecognised in patients with inflammatory bowel disease.

The SeHCAT (seleno-tauro-homocholic acid) test is currently the only diagnostic test for BAM, but it is not widely available and it is also time consuming, expensive and involves exposure to radioactivity. Some clinicians give a course of blind or empirical treatment instead. The National Institute of Clinical Excellence (NICE) recognised these issues and highlighted the need for cheaper and safer tests to identify BAM.

This study will assess the accuracy of a simple, convenient and inexpensive laboratory test for the rapid diagnosis of BAM which measures bile acids in stool. This test has the potential to have a broad impact on clinical practice and patient care by enabling doctors to identify and treat patients with BAM promptly. Results from the second phase of the study will allow the assessment of the benefits of monitoring the stool test to determine whether the bile acid changes can predict the response to treatment and dosage needed for each patient.

DETAILED DESCRIPTION:
The prevalence of chronic diarrhoea is 5% of the population, a third of these cases have bile acid malabsorption (BAM).

SeHCAT (seleno-tauro-homocholic acid) testing is the gold standard for BAM, and involves the ingestion of seleno-tauro-homocholic acid, which is limited to a small number of UK centres. NICE reported that although SeHCAT might benefits patients, there was a need to explore alternative technologies.

With limited access to and cost of SeHCAT, many centres use an empirical trial of bile acid sequestrants, without a diagnosis. This may not be effective as many patients are non-adherent.

This pilot study will evaluate a cheaper and simpler laboratory test, which quantitates faecal bile acids. This assay is safer, easier to use, and potentially gives a rapid diagnosis in BAM. The aim is to determine the sensitivity and specificity of this new assay. In the longitudinal phase of this study, further evaluate of faecal bile acids following bile salt sequestrant therapy, will evaluate its role in dose titration.

The following patients will be recruited (i) post-cholecystectomy; (ii) post-terminal ileal resection; or (iii) primary BAM. Patients will have SeHCAT testing and the faecal bile acid concentration will be determined.

Outcomes: The results of faecal bile acid measurement in these patients will be compared with SeHCAT to determine its sensitivity and specificity. Longitudinal follow up will determine the effect of bile salt sequestration on faecal bile acids. These results would inform the design of larger studies, allowing the evaluation of this new test in the NHS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years age and over
* Willing to provide informed consent
* Post-cholecystectomy patients group (n=30; type 3 BAD)
* Post-terminal ileal resection patients with Crohn's disease group (n=30; type 1 BAD)
* D-IBS patients with normal SeHCAT retention group (n=30)
* Idiopathic bile salt diarrhoea with abnormal SeHCAT retention group (type 2 BAD) (n=30)

Exclusion Criteria:

* Pregnancy/ breast feeding
* Patient participating in another trial
* Patients unable to give written consent
* Known established bile salt diarrhoea
* Recipients of antibiotics in under 4 weeks of initial trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
faecal bile acids retention values. | 12 weeks
SeHCAT retention values | 12 weeks

SECONDARY OUTCOMES:
measurement of faecal bile acids | 12 weeks
  Sensitivity and specificity of positive and negative predictive values
measurement of bile salt sequestrants | 12 weeks
  descriptive prediction on the response to treatment
excretion of faecal bile acids | 12 weeks
  descriptive prediction on the response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A single faecal bile acid stool test demonstrates potential efficacy in replacing SeHCAT testing for bile acid diarrhoea in selected patients — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9117305/
- See also: The impact of bile acid sequestrants on quality of life in patients with bile acid diarrhoea. — https://pubmed.ncbi.nlm.nih.gov/35778677/
- See also: Pre-analytical DNA yield and variability influences microbiome laboratory analyses: is it time for a unified international consensus for optimal sampling and DNA isolation? — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9223004/
- See also: The analysis of gut microbiota in patients with bile acid diarrhoea treated with colesevelam. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10063896/
- See also: Bile acids and the gut microbiome in post-operative Crohn's disease: a mechanistic relationship? — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8964223/